CLINICAL TRIAL: NCT02143401
Title: A Phase I Trial of ABT-263 (Navitoclax), a Bcl-2 Inhibitor, and Sorafenib (Nexavar) in Patients With Relapsed or Refractory Solid Organ Tumors
Brief Title: Navitoclax and Sorafenib Tosylate in Treating Patients With Relapsed or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-01043; NCI-2014-01043 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1315; 9608 (Other: Mayo Clinic Cancer Center LAO); 9608 (Other: CTEP); UM1CA186686 (NIH)
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Cirrhosis; Hepatitis B Infection; Hepatitis C Infection; Metastatic Malignant Solid Neoplasm; Recurrent Hepatocellular Carcinoma; Recurrent Malignant Solid Neoplasm; Refractory Malignant Neoplasm; Stage IV Hepatocellular Carcinoma AJCC v7; Unresectable Solid Neoplasm
MeSH Terms: conditions — Fibrosis; Hepatitis B; Hepatitis C; Neoplasm Metastasis; Carcinoma, Hepatocellular; Neoplasms | interventions — navitoclax; Sorafenib

ARMS (1):
- Treatment (navitoclax, sorafenib tosylate) (Experimental): Patients receive navitoclax PO QD on days 1-21 (days 1-28 cycle of 1 only) and sorafenib tosylate PO BID on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Navitoclax; Other: Pharmacological Study; Drug: Sorafenib; Drug: Sorafenib Tosylate

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Navitoclax — Given PO
  Other Names: A-855071.0; ABT-263; BcI-2 Family Protein Inhibitor ABT-263
Other: Pharmacological Study — Correlative studies
Drug: Sorafenib — Given PO
  Other Names: BA4 43 9006; BAY 43 9006; BAY 43-9006; BAY 439006; BAY-43-9006; Bay-439006; BAY439006
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54 9085; BAY 54-9085; BAY 549085; BAY-54-9085; BAY549085; Nexavar; sorafenib

SUMMARY:
This phase I trial studies the side effects and the best dose of navitoclax when given together with sorafenib tosylate in treating patients with solid tumors that have returned (relapsed) or do not respond to treatment (refractory). Navitoclax and sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of the combination of navitoclax and sorafenib tosylate (sorafenib) in patients with advanced solid tumors. (Dose escalation cohort) II. To better characterize the toxicity profile of the combination of navitoclax and sorafenib. (Dose expansion cohort)

SECONDARY OBJECTIVES:

I. To identify any activity of this treatment combination in patients with metastatic cancer. (Dose escalation cohort) II. To seek preliminary evidence of activity of this treatment combination in patients with hepatoma. (Dose expansion cohort)

CORRELATIVE OBJECTIVES:

I. To determine whether the combination of navitoclax and sorafenib induces apoptosis that can be detected by peripheral blood biomarker analysis. (Dose escalation cohort) II. To assess peripheral blood biomarkers and pharmacokinetics in a more homogenous population. (Dose expansion cohort) III. To determine whether treatment is associated with Mcl-1 down regulation in hepatocellular carcinoma (HCC) at the maximum tolerated dose (MTD). (Dose expansion cohort) IV. To assess in a preliminary fashion whether pretreatment tumor cell levels of Mcl-1 predict response to this regimen through serial biopsies. (Dose expansion cohort)

OUTLINE: This is a dose-escalation study of navitoclax.

Patients receive navitoclax orally (PO) once daily (QD) on days 1-21 (days 1-28 cycle of 1 only) and sorafenib tosylate PO twice daily (BID) on days 1-21. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* For Dose Escalation Cohort: Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* For Dose Expansion Cohort: HCC patients only: HCC confirmed by biopsy OR diagnosed by clinical and radiologic criteria; all of the following criteria must be met or a biopsy is required:

  * Known cirrhosis or chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
  * Hypervascular liver masses > 2 cm, and either serum alpha-fetoprotein (AFP) > 400 ng/ml
  * AFP > three times normal and doubling in value in the antecedent 3 months
  * In the expansion cohort, prior treatment with sorafenib as first-line therapy allowed
* Any number of the following prior therapies is allowed:

  * Chemotherapy >= 28 days prior to registration
  * Mitomycin C/nitrosoureas >= 42 days prior to registration
  * Immunotherapy >= 28 days prior to registration
  * Biologic therapy >= 28 days prior to registration
  * Targeted therapy >= 28 days prior to registration
  * Radiation therapy >= 28 days prior to registration
  * Radiation to < 25% of bone marrow
* HCC patients only: Prior regional treatments for liver metastasis are permitted including:

  * Selective internal radiation therapy such as brachytherapy, cyber knife, radiolabeled microsphere embolization, etc.
  * Hepatic artery chemoembolization
  * Hepatic artery embolization
  * Hepatic artery infusional chemotherapy
  * Radiofrequency ablation
  * NOTE: patients must be >= 4 weeks from treatment and show progressive measurable/evaluable disease in the liver after regional therapy or must have measurable disease outside the liver
* HCC patients only: Child Pugh class A or B7 liver disease
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Life expectancy of > 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL (patients may be treated with hematopoietic growth factors to achieve or maintain this level)
* Hemoglobin >= 9.0 g/dL
* International normalized ratio (INR) =< 1.4
* Platelets >= 100,000/mm^3
* Total bilirubin =< 1.5 x ULN (institutional upper limit of normal) (patients with Gilbert's syndrome may have direct bilirubin > 2.5 x ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN
* Serum creatinine =< 1.5 x ULN
* Able to swallow and retain oral medication
* Negative serum pregnancy test =< 7 days prior to registration for women of childbearing potential

  * NOTE: women will be considered not of childbearing potential if they are surgically sterile (bilateral oophorectomy or hysterectomy) and/or post-menopausal (amenorrheic for at least 12 months)
* Ability to understand and the willingness to sign a written informed consent document
* Willing to provide tissue samples for correlative research purposes

Exclusion Criteria:

* Unresolved toxicity of National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (NCI CTCAE v 4.0) grade 2 or higher from previous anti-cancer therapy, except alopecia
* Receiving any other investigational agents =< 28 days prior to registration
* Known brain metastases (even if treated)
* Known portal hypertension or history of variceal bleeding; these patients are felt to be at increased risk of bleeding if they experience navitoclax-induced thrombocytopenia
* Inadequately controlled hypertension (systolic blood pressure of > 150 mmHg or diastolic pressure > 90 mmHg on anti-hypertensive medications)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to navitoclax or sorafenib
* Current use of anticoagulation; NOTE: use of low-dose anticoagulation medications that are used to maintain the patency of a central intravenous catheter is allowed
* Corrected QT (QTc) interval > 480 msec on baseline electrocardiogram (EKG)
* Documented history of prolonged QTc interval =< 6 months prior to registration
* Receiving any medications that prolong the QTc and have a known risk for Torsades de pointes; providers should use caution with drugs with possible increased risk for Torsades de pointes; NOTE: patient will be eligible if they can be taken off these medications prior to initiation of therapy and no less than 4 half-lives of the medication
* Current use of certain concomitant medications due to mechanistic-based platelet toxicities from navitoclax: clopidogrel, ibuprofen, tirofiban and other anticoagulants, drugs or herbal supplements that effect platelet function; NOTE: antiplatelet use is prohibited during the use of navitoclax; subjects who have previously received aspirin therapy for thrombosis prevention may resume a low dose (i.e., maximum 100 mg QD) of aspirin if platelet counts are stable (>= 50,000/mm^3) through 6 weeks of navitoclax administration; all decisions regarding treatment with aspirin therapy will be determined by the principal investigator in conjunction with the medical monitor
* Current use of strong CYP3A inhibitors such as ketoconazole, itraconazole, voriconazole, posaconazole, nefazodone, and clarithromycin are prohibited; NOTE: moderate inhibitors of CYP3A4 should be used with caution; navitoclax is a moderate inhibitor of CYP2C8 and a strong inhibitor of CYP2C9; caution should be exercised when dosing navitoclax concurrently with CYP2C8 and CYP2C9 substrates; common CYP2C8 substrates include paclitaxel, statins and repaglinide; CYP2C9 substrates include celecoxib, phenytoin and warfarin; when possible, investigators should switch to alternative medications or monitor the patients closely
* Concurrent use of strong CYP3A4/5 inducers such as carbamazepine, phenytoin, rifampin, and St. John's wort are prohibited
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any of the following:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential who are unwilling to employ adequate contraception; NOTE: should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; the effects of navitoclax on the developing human fetus are unknown; for this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception using one of the methods listed below prior to study entry, for the duration of study participation, and up to 90 days following completion of therapy:

    * Total abstinence from sexual intercourse (minimum one complete menstrual cycle prior to study drug administration)
    * Vasectomized male subject or vasectomized partner of female subjects
    * Hormonal contraceptives (oral, parenteral, transdermal or vaginal ring) for at least 3 months prior to study drug administration; if the subject is currently using a hormonal contraceptive, she should also use a barrier method during this study and for 1 month after study completion
    * Intrauterine device (IUD)
    * Double-barrier method: male condom plus diaphragm or vaginal cap with spermicide (contraceptive sponge, jellies or creams)
    * Additionally, male subjects (including those who are vasectomized) whose partners are pregnant or might be pregnant must agree to use condoms for the duration of the study and for 90 days following completion of therapy
* Human immunodeficiency virus (HIV)-positive patients on highly active antiretroviral therapy (HAART) are excluded due to possible drug-drug interactions with the investigational agent(s)
* Underlying condition predisposing them to bleeding or currently exhibits signs of clinically significant bleeding
* Recent history of non-chemotherapy-induced thrombocytopenic-associated bleeding =< 1 year prior to the registration
* History of cardiovascular disease (e.g., myocardial infraction [MI], thrombotic or thromboembolic event in the last 6 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-01-30 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of navitoclax | 28 days
  Will be defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients) per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 4.0.
Incidence of adverse events | Up to 3 months
  Will be graded per NCI CTCAE v. 4.0. The number and severity of all adverse events (overall, by dose-level, and by tumor group) will be tabulated and summarized in this patient population. The grade 3+ adverse events will also be described and summarized in a similar fashion.

SECONDARY OUTCOMES:
Tumor response | Up to 3 months
  Will be assessed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline version 1.1. Response will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease. The waterfall plot may be used to display best tumor response. Exploratory analysis of the relationship between response and other clinical endpoints may be performed.
Time until any treatment related toxicity | Up to 3 months
  The data on time-related variables will be summarized descriptively.
Time until treatment related grade 3+ toxicity | Up to 3 months
  The data on time-related variables will be summarized descriptively.
Time until hematologic nadirs (white blood cell, absolute neutrophil count, platelets) | Up to 3 months
  The data on time-related variables will be summarized descriptively.
Time to progression | Up to 3 months
  The data on time-related variables will be summarized descriptively.
Time to treatment failure | From registration to documentation of progression, unacceptable toxicity, or refusal to continue participation by the patient, assessed up to 3 months
  The data on time-related variables will be summarized descriptively.

OTHER OUTCOMES:
Changes in levels of cleaved cytokeratin 18 (expansion cohort only) | Day -7 up to day 8
  To assess changes in each antigen, dot plots will be constructed with H-score on the Y axis and pre-or post-treatment status on the X axis, looking for patterns of change that emerge. To assess whether changes occur predominantly in one direction, a sign test will be applied.
Changes in hepatoma Mcl-1 expression level in tumor tissue (expansion cohort only) | Baseline to up to day 8
  Will be assessed by immunohistochemistry. The relationship between pretreatment Mcl-1 expression and clinical response will be examined in a post hoc and exploratory fashion. To assess the relationship between Mcl-1 and response the H score (0-300) vs. response will be graphed. Chi-squared tests will be used to assess significance of relationships between these dichotomous variables and response. In addition, associations between molecular markers and time-to-event variables (progression-free-survival [PFS]) will be illustrated graphically using Kaplan-Meier curves and log-rank tests in an exploratory fashion.
Change in cleaved and total CK18 levels in serum | Day -7 to up to day 8
  Will be assessed by enzyme-linked immunosorbent assay (ELISA). Will be summarized descriptively and plotted along time by dose levels and as a whole. The changes of the serum levels of cleaved and total CK18 at each time point against pre-treatment baseline will be correlated with toxicity and clinical endpoints. The relationships between cleaved and total CK18, caspase 3 and cytochrome c at various time points and dose levels will be explored in longitudinal data analysis. Tissue expression of Mcl-1 will be correlated with serum levels of cleaved and total CK18 at different time points and clinical toxicity and tumor response.

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Costello, Principal Investigator — Mayo Clinic Cancer Center LAO
Locations (10):
- United States (10):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas